CLINICAL TRIAL: NCT06799962
Title: Assistance and Rehabilitation of Eating Behavior Through Devices Based on Artificial Intelligence and Virtual Reality
Brief Title: AI and VR Devices for Eating Behavior Rehabilitation
Acronym: ARCADIA-VR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Collaborators: Madre Teresa s.r.l (Unknown); Medilink s.r.l. (Unknown); SB SETEC S.p.A (Unknown); Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Flavia Marino, Head of Unit, Istituto per la Ricerca e l'Innovazione Biomedica
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CNR-IRIB-PRO-2025-001
Record Dates: First submitted 2025-01-24; First posted 2025-01-29 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Eating Disorders; Anorexia Nervosa; Bulimia Nervosa
Keywords: Eating Disorders; Anorexia Nervosa; Bulimia Nervosa; Virtual Reality; Artificial Intelligence; Body Perception; Emotional Regulation; Cognitive Behavioral Therapy
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa; Bulimia Nervosa; Emotional Regulation | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Intervention Group for Anorexia Nervosa (Experimental): Participants diagnosed with Anorexia Nervosa will undergo treatment enhanced with Virtual Reality (VR) and Artificial Intelligence (AI) technologies, specifically the Enhanced Body-Swap system. The intervention targets body perception and emotional regulation to address symptoms and improve treatment outcomes.
  Interventions: Other: Enhanced Body-Swap for Anorexia Nervosa
- Intervention Group for Bulimia Nervosa (Experimental): Participants diagnosed with Bulimia Nervosa will receive treatment incorporating VR and AI technologies, specifically the Emotional Rescripting system. The intervention aims to modify emotional experiences and cognitive responses associated with binge-purge behaviors.
  Interventions: Other: Emotional Rescripting for Bulimia Nervosa
- Control Group for Anorexia Nervosa (Other): Participants diagnosed with Anorexia Nervosa will follow the same therapeutic protocol as ARM 1 but without the integration of VR and AI technologies. This group serves as a comparison to assess the added value of VR and AI in treatment.
  Interventions: Other: Standard Therapy for Anorexia Nervosa (Control)
- Control Group for Bulimia Nervosa (Other): Participants diagnosed with Bulimia Nervosa will follow the same therapeutic protocol as ARM 2 but without the inclusion of VR and AI technologies. This group serves as a baseline to evaluate the impact of VR and AI in treatment.
  Interventions: Other: Standard Therapy for Bulimia Nervosa (Control)

INTERVENTIONS:
Other: Enhanced Body-Swap for Anorexia Nervosa — The protocol begins with a baseline session, where participants familiarize themselves with their virtual body and provide anamnesis and therapeutic efficacy baseline data. The treatment phase includes 12 bi-weekly sessions where participants embody a virtual avatar in a VR environment. During each session, the Body Mass Index (BMI) of the virtual body is incrementally increased toward a target BMI approximating normal weight (18.5). Follow-ups are conducted at 4, 8, and 12 weeks to assess long-term effects.
  Arms: Intervention Group for Anorexia Nervosa
Other: Emotional Rescripting for Bulimia Nervosa — The protocol starts with an assessment phase (1 session), gathering anamnesis and baseline therapeutic efficacy data. This is followed by an evaluation phase (2 sessions), where participants rate craving responses for virtual foods and environments in immersive VR, with physiological data collected via biosensors. Using this data, a personalized exposure hierarchy is created, combining the most craving-inducing foods and environments into 40 interactive 3D scenarios. The treatment phase involves 9 VR sessions focusing on emotional regulation and craving management. Follow-ups at 4, 8, and 12 weeks evaluate progress.
  Arms: Intervention Group for Bulimia Nervosa
Other: Standard Therapy for Anorexia Nervosa (Control) — Participants follow a similar structure with a baseline session to collect anamnesis and baseline data, but without VR immersion. The treatment phase consists of 12 bi-weekly sessions of standard cognitive-behavioral therapy (CBT), focusing on addressing maladaptive thought patterns, promoting healthy eating behaviors, and reducing body image disturbances. Follow-ups are conducted at 4, 8, and 12 weeks to monitor progress. No VR or AI technologies are integrated.
  Arms: Control Group for Anorexia Nervosa
Other: Standard Therapy for Bulimia Nervosa (Control) — Participants undergo an assessment phase (1 session) to collect baseline data and an evaluation phase (2 sessions) using standard craving questionnaires without VR immersion or biosensors. The treatment phase includes 9 sessions of traditional CBT targeting binge-purge cycles and emotional triggers. Follow-ups at 4, 8, and 12 weeks monitor progress without the integration of VR or AI technologies.
  Arms: Control Group for Bulimia Nervosa

SUMMARY:
Eating disorders (ED) affect the relationship with food and body image. Virtual reality (VR), combined with artificial intelligence (AI), offers new clinical solutions, overcoming traditional cognitive behavioral therapy (CBT). The ARCADIA VR project aims to develop devices to treat ED through personalized VR systems (e.g. Enhanced Body-Swap for anorexia, Emotional Rescripting for bulimia) and AI predictive algorithms to monitor severity, risk and efficacy of treatments. These approaches promise better and faster results, improving diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Anorexia Nervosa or Bulimia Nervosa according to DSM-5-TR (APA, 2013) and ICD-11, confirmed by a public hospital setting
* Body Mass Index (BMI) between 16 and 32
* Disorder present for at least 6 months
* No other concurrent psychotherapeutic interventions during the study
* All participants with a previous diagnosis will be re-evaluated and confirmed through assessment and consent by expert professionals in the research team (i.e., a neuropsychiatrist and a clinical psychologist)

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Eating Disorder Inventory-3 (EDI-3) | For Bulimia Nervosa the evaluations will be at T0 (baseline),T1 (monitoring at 5 weeks), T2 (post-intervention at 9 weeks), and T3 (follow-up at 12 weeks). For Anorexia Nervosa will be at T0 (baseline), 5 weeks (T1), 9 weeks (T2), and 12 weeks (T3)
  The EDI-3 is a standardized self-report questionnaire widely used to assess symptoms and psychological traits associated with the development and maintenance of eating disorders. It includes 91 items across 12 scales, using a 6-point Likert scale ranging from 0 (never) to 5 (always).
Physical Appearance State and Trait Anxiety Scale (PASTAS) | For Anorexia Nervosa the evaluation sessions will be scheduled at T0 (baseline), 5 weeks (T1), 9 weeks (T2), and 12 weeks (T3) and will last 5 minutes.
  The PASTAS is a validated measure for assessing state and trait anxiety related to body image. Participants rate their anxiety and nervousness about their physical appearance, including negative thoughts and physiological responses, on a 5-point Likert scale (0 = never, 5 = always)
Body Image Assessment Scale-Body Dimensions (BIAS-BD) | For Anorexia Nervosa, the evaluation sessions will be scheduled at T0 (baseline), 5 weeks (T1), 9 weeks (T2), and 12 weeks (T3) and will last 15 minutes.
  The BIAS-BD evaluates the perceptual and emotional components of body image dimensions. It measures the discrepancy between perceived and ideal body size (body dissatisfaction) and the discrepancy between perceived and actual body size (body distortion). It uses a range of 17 silhouettes, with different versions for males and females.
Body Appreciation Scale-2 (BAS-2) | For Anorexia Nervosa, the evaluation sessions will be scheduled at T0 (baseline), 5 weeks (T1), 9 weeks (T2), and 12 weeks (T3) and will last 10 minutes.
  The BAS-2 is a 10-item measure that assesses body appreciation. Participants rate statements on a 5-point Likert scale (1 = never, 5 = always). Higher scores indicate greater body appreciation. Example items include "I respect my body" and "I feel comfortable in my body."
Objectified Body Consciousness Scale (OBCS) | For Anorexia Nervosa the evaluation sessions will be scheduled at T0 (baseline), 5 weeks (T1), 9 weeks (T2), and 12 weeks (T3) and will last 10 minutes.
  The OBCS consists of 24 items grouped into three subscales: body control, body shame, and appearance control beliefs. Each subscale includes 8 items rated on a 7-point Likert scale (1 = strongly disagree, 7 = strongly agree). Subscale scores are calculated as means, with higher scores indicating greater levels of the measured variable.
Body Uneasiness Test (BUT) | For Anorexia Nervosa the evaluation sessions will be scheduled at T0 (baseline), 5 weeks (T1), 9 weeks (T2), and 12 weeks (T3) and will last 10 minutes.
  The BUT is a 34-item self-report questionnaire focusing on body dissatisfaction and body-related emotions such as anxiety, concern, and embarrassment. It comprises five subscales-weight phobia, body image concern, avoidance, compulsive self-monitoring, and depersonalization-and a general score. This tool is validated in Italian.
Food Craving Questionnaire (FCQ) | For Bulimia Nervosa the evaluation session will be divided into three moments and will last 15 minutes. The proposed evaluation moments are T0 (baseline), T1 (monitoring at 5 weeks), T2 (post-intervention at 9 weeks), and T3 (follow-up at 12 weeks).
  The FCQ measures the intensity of food cravings both as a trait (habitual experiences) and as a state (current experiences). The FCQ-Trait comprises 39 items rated on a 6-point Likert scale (never to always), while the FCQ-State comprises 15 items rated on a 5-point Likert scale (1 = strongly disagree, 5 = strongly agree).
Binge Eating Scale (BES) | For Bulimia Nervosa the evaluation session will be divided into three moments and will last 5 minutes. The proposed evaluation moments are T0 (baseline), T1 (monitoring at 5 weeks), T2 (post-intervention at 9 weeks), and T3 (follow-up at 12 weeks).
  The BES is a self-report tool designed to identify and quantify the severity of Binge Eating Disorder (BED). It assesses the frequency of binge episodes, associated behaviors, and emotional experiences during and after binge eating. Higher scores indicate greater severity of BED symptoms.
Difficulties in Emotional Regulation Scale (DERS-20) | For Bulimia Nervosa the evaluation session will be divided into three moments and will last 10 minutes. The proposed evaluation moments are T0 (baseline), T1 (monitoring at 5 weeks), T2 (post-intervention at 9 weeks), and T3 (follow-up at 12 weeks).
  The DERS is a self-report questionnaire assessing emotional regulation abilities. The Italian short version (DERS-20) includes 20 items rated on a 5-point Likert scale (1 = almost never, 5 = almost always) and measures five dimensions: lack of acceptance, difficulty engaging in goal-directed behavior, lack of control, difficulty recognizing emotions, and reduced self-awareness. Higher scores indicate greater difficulties in emotional regulation.
State and Trait Anxiety Inventory (STAI) | For Bulimia Nervosa the evaluation session will be divided into three moments and will last 20 minutes. The proposed evaluation moments are T0 (baseline), T1 (monitoring at 5 weeks), T2 (post-intervention at 9 weeks), and T3 (follow-up at 12 weeks).
  The STAI is a self-report questionnaire measuring state anxiety (temporary condition) and trait anxiety (long-standing tendency). It consists of 40 items rated on a 4-point Likert scale (almost never to almost always). Twenty items assess state anxiety (STAI-S), and 20 assess trait anxiety (STAI-T). Higher scores indicate higher levels of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Flavia Marino, Principal Investigator — Institute for Biomedical Research and Innovation (IRIB) - National Research Council (CNR)
Locations (1):
- Institute for Biomedical Research and Innovation (IRIB) - National Research Council (CNR), Messina, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brown T, Nauman Vogel E, Adler S, Bohon C, Bullock K, Nameth K, Riva G, Safer DL, Runfola CD. Bringing Virtual Reality From Clinical Trials to Clinical Practice for the Treatment of Eating Disorders: An Example Using Virtual Reality Cue Exposure Therapy. J Med Internet Res. 2020 Apr 23;22(4):e16386. doi: 10.2196/16386. PMID 32324145
- [Background] Demartini B, Goeta D, Romito L, Anselmetti S, Bertelli S, D'Agostino A, Gambini O. Anorexia Nervosa and Functional Motor Symptoms: Two Faces of the Same Coin? J Neuropsychiatry Clin Neurosci. 2017 Fall;29(4):383-390. doi: 10.1176/appi.neuropsych.16080156. Epub 2017 May 31. PMID 28558480
- [Background] Colombo D, Diaz-Garcia A, Fernandez-Alvarez J, Botella C. Virtual reality for the enhancement of emotion regulation. Clin Psychol Psychother. 2021 May;28(3):519-537. doi: 10.1002/cpp.2618. Epub 2021 Jun 23. PMID 34048621
- [Background] Clus D, Larsen ME, Lemey C, Berrouiguet S. The Use of Virtual Reality in Patients with Eating Disorders: Systematic Review. J Med Internet Res. 2018 Apr 27;20(4):e157. doi: 10.2196/jmir.7898. PMID 29703715
- [Background] Boeldt D, McMahon E, McFaul M, Greenleaf W. Using Virtual Reality Exposure Therapy to Enhance Treatment of Anxiety Disorders: Identifying Areas of Clinical Adoption and Potential Obstacles. Front Psychiatry. 2019 Oct 25;10:773. doi: 10.3389/fpsyt.2019.00773. eCollection 2019. PMID 31708821
- [Background] Badoud D, Tsakiris M. From the body's viscera to the body's image: Is there a link between interoception and body image concerns? Neurosci Biobehav Rev. 2017 Jun;77:237-246. doi: 10.1016/j.neubiorev.2017.03.017. Epub 2017 Apr 1. PMID 28377099